CLINICAL TRIAL: NCT00762996
Title: The Clinical Evaluation of Two Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Eurolens Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0707
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2009-06-23 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- etafilcon A/etafilcon A (Active Comparator): Period 1: etafilcon A, Period 2: etafilcon A
  Interventions: Device: etafilcon A
- etafilcon A/omafilcon A (Active Comparator): Period 1: etafilcon A, Period 2: omafilcon A
  Interventions: Device: etafilcon A; Device: omafilcon A
- omafilcon A/etafilcon A (Active Comparator): Period 1: omafilcon A, Period 2: etafilcon A
  Interventions: Device: etafilcon A; Device: omafilcon A
- omafilcon A/omafilcon A (Active Comparator): Period 1: omafilcon A, Period 2: omafilcon A
  Interventions: Device: omafilcon A

INTERVENTIONS:
Device: etafilcon A — contact lens
  Arms: etafilcon A/etafilcon A; etafilcon A/omafilcon A; omafilcon A/etafilcon A
Device: omafilcon A — contact lens
  Arms: etafilcon A/omafilcon A; omafilcon A/etafilcon A; omafilcon A/omafilcon A

SUMMARY:
The objective of this study is to evaluate the clinical performance of two daily disposable contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* They are of legal age (18 years) and capacity to volunteer.
* They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
* They are willing and able to follow the protocol.
* They would be expected to attain at least 6.9 (20/30) in each eye with the study lenses.
* They are able to wear contact lenses which have a back vertex power of -1.00 to -6.00DS.
* They have a maximum of 1.00D of refractive astigmatism (i.e. < 1.00 DC).
* They have worn soft contact lenses within six months of starting the study.

Exclusion Criteria:

* They have an ocular disorder which would normally contra-indicate contact lens wear.
* They have a systemic disorder which would normally contra-indicate contact lens wear.
* They are using any topical medication such as eye drops or ointment.
* They are aphakic.
* They have had corneal refractive surgery.
* They have any corneal distortion resulting from previous hard or rigid lens wear or has keratoconus.
* They are pregnant or lactating.
* They have grade 2 or greater of any of the following ocular surface signs: corneal edema, corneal vascularization, corneal staining, tarsal conjunctival changes or any other abnormality which would normally contraindicate contact lens wear.
* They have any infectious disease (e.g., hepatitis) or any immunosuppressive disease (e.g., HIV).
* They have diabetes.
* They are currently taking part in any other clinical study or research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Etafilcon A / Etafilcon A: Period 1: etafilcon A, Period 2: etafilcon A
- Etafilcon A / Omafilcon A: Period 1: etafilcon A, Period 2: omafilcon A
- Omafilcon A / Etafilcon A: Period 1: omafilcon A, Period 2: etafilcon A
- Omafilcon A / Omafilcon A: Period 1: omafilcon A, Period 2: omafilcon A
Period: Period One
Arm/Group | Etafilcon A / Etafilcon A | Etafilcon A / Omafilcon A | Omafilcon A / Etafilcon A | Omafilcon A / Omafilcon A
Started | 15 | 16 | 17 | 17
Completed | 15 | 16 | 13 | 16
Not Completed | 0 | 0 | 4 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — ineligible | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Period: Period Two
Arm/Group | Etafilcon A / Etafilcon A | Etafilcon A / Omafilcon A | Omafilcon A / Etafilcon A | Omafilcon A / Omafilcon A
Started | 15 | 16 | 13 | 16
Completed | 15 | 16 | 13 | 16
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Population
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity
Description: logarithm of the minimum angle of resolution (logMar) ideal is 0.0 and represents 20/20 Snellen acuity. logMar values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal.
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: logMar
Arm/Group | Etafilcon A | Omafilcon A
Number analyzed (Participants) | 44 | 45
logMar | 0.03460 (0.007129) | 0.02931 (0.006666)
Statistical Analysis 1: Comparison: Etafilcon A vs Omafilcon A; Null Hypothesis: etafilcon A is greater than or equal to omafilcon A; Test type: Non-Inferiority or Equivalence — margin +/- 0.5 logMar lines The range of non-inferiority for this value is 0.50 thus +/- 0.50 is considered non-inferior to the 0.0 mark. logarithm of the minimum angle of resolution (logMar) ideal is 0.0 and represents 20/20 Snellen acuity. logMar values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal; Mixed Models Analysis; Mean Difference (Final Values) = 0.005287, 95% CI [-0.01389 to 0.2447], Standard Error of Mean 0.009760 — logarithm of the minimum angle of resolution (logMar) ideal is 0.0 and represents 20/20 Snellen acuity. logMar values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal

2. Secondary Outcome: Lens Comfort
Description: A weighted combined score calculated from individual comfort-related questions asked on a 1-5 scale: 1=most negative response to 5=most positive was used to derive comfort outcomes. The analysis shows the difference in outcome between the test and control.>0 = comfortable, <0 = uncomfortable
Time Frame: 1 week
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Etafilcon A | Omafilcon A
Number analyzed (Participants) | 15 | 16
Units on a scale | 0.3113 (0.1765) | -0.1645 (0.2075)
Statistical Analysis 1: Comparison: Etafilcon A vs Omafilcon A; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.4757, 95% CI [0.05563 to 0.4757], Standard Error of Mean 0.2505 — Mean difference is etafilcon A minus omafilcon A

ADVERSE EVENTS:
Arm/Group | Etafilcon A / Etafilcon A | Etafilcon A / Omafilcon A | Omafilcon A / Etafilcon A | Omafilcon A / Omafilcon A
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/10 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/15 | 0/10 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.